CLINICAL TRIAL: NCT06555575
Title: A Randomized Controlled Trial of Ubiquinone vs Ubiquinol Supplementation in Women Over Age 37 Undergoing in Vitro Fertilization.
Brief Title: Ubiquinone vs. Ubiquinol Supplementation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Trio Fertility (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K001
Record Dates: First submitted 2024-08-08; First posted 2024-08-15 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: IVF
Keywords: ubiquinone; ubiquinol; reproductive outcome
MeSH Terms: interventions — Ubiquinone; ubiquinol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- coQ10 A (Experimental): Eligible subjects will be receiving ubiquinone 200 mg prior to their in vitro fertilization (IVF) cycle.
  Interventions: Drug: Ubiquinone 200 Mg Oral Capsule
- coQ10B (Experimental): Eligible subjects will be receiving ubiquinol 100 mg prior to their IVF cycle.
  Interventions: Drug: Ubiquinol 100 MG Oral Capsule
- Control (No Intervention): Subjects are not receiving coQ10 supplementation.

INTERVENTIONS:
Drug: Ubiquinone 200 Mg Oral Capsule — By mouth three times daily for three months
  Arms: coQ10 A
Drug: Ubiquinol 100 MG Oral Capsule — By mouth three times daily for three months
  Arms: coQ10B

SUMMARY:
The objective of this study is to determine if ubiquinol will result in improved reproductive outcomes in older women at a reduced oral dose compared to current standard treatment with ubiquinone.

DETAILED DESCRIPTION:
As more women choose to delay child rearing, it has become increasingly important to understand why fertility declines with increasing maternal age. One of the factors suggested to play a role in reproductive aging is mitochondrial aging. Mitochondria are considered to be the batteries of the eggs and are responsible for generating energy necessary for egg and subsequent embryo development.

The egg maturation process involves a combination of many changes - all of which require energy that is provided by the mitochondria. Coenzyme Q10 (CoQ10) plays an important role as fuel in this process.

The investigators have shown that CoQ10 is needed for proper energy production by mitochondria and its addition to the diet could act as a potential treatment for egg aging.

It has been shown that in an aged mouse model, administration of CoQ10 (ubiquinone) results in improved mitochondrial energy production, more healthy embryos and more live-born pups. In clinical studies, the investigators also showed potential beneficial effects to increase the number of normal embryos from human eggs in older patients. So far, only one small study measured CoQ10 concentrations in the fluid that surrounds the eggs inside the ovaries (follicular fluid) and found significantly higher CoQ10 in the follicular fluid of normal mature eggs vs abnormal eggs. In addition, higher CoQ10 concentrations were also associated with better quality embryos. This study supports the hypothesis that CoQ10 supplementation may improve egg and embryo quality.

So far, all the research studies of CoQ10 in reproductive aging have administered a form of CoQ10 called ubiquinone. Another form of CoQ10 (ubiquinol), appears to be absorbed by the body better than ubiquinone and may have other beneficial effects in the ovary besides just increasing energy production.

ELIGIBILITY:
Inclusion Criteria:

1. Women age >37 and <43 years undergoing their first in vitro fertilization (IVF) cycle
2. Day 3 follicle-stimulating hormone (FSH) <12 IU/L with serum estradiol <250 pmol/L and normal thyroid-stimulating hormone (TSH) and Prolactin
3. Partner with semen analysis suitable for IVF or ICSI
4. Anti-müllerian hormone (AMH) > 3 pmol/L
5. Be willing and able to provide written informed consent for the study.
6. Be an otherwise healthy female and considered eligible by the investigator to be treated with a daily dose of 225 IU Recombinant human FSH (recFSH) and 75 IU Human menopausal gonadotrophins (hMG).
7. Documented history of infertility for at least 12 months before randomization (not applicable in case of tubal infertility or severe male factor infertility, or when the use of donor sperm is indicated)
8. Have a body mass index (BMI) ≥17.5 and ≤38 kg/m2
9. Have available ejaculatory sperm (use of donated and/or cryopreserved sperm is allowed)
10. Have a normal uterine cavity (no evidence of uterine polyp or submucosal fibroid) as assessed by either saline-infused sonohysterography or by hysteroscopy within 12 months of randomization
11. Have results of clinical laboratory tests (hematology, serum chemistry, and urinalysis) within normal limits or clinically acceptable to the investigator
12. Has a pelvic ultrasound showing no cyst ≥15 mm

Exclusion Criteria:

1. Has been diagnosed with or treated for any endocrine abnormality within 3 years prior Note: Participants with a history of clinical or subclinical hypothyroidism may be eligible if thyroid stimulating hormone levels at screening are within normal limits and the participant has been on a stable dose of thyroid replacement medication (or on no replacement therapy) for at least 8 weeks.
2. Has a prolactin level above the upper limit of normal for the central laboratory
3. Has FSH >12.0 IU/L
4. Has a history of a full or partial resection of an ovary, including a history of ovarian cystectomy, or of any ovarian tumors limiting access to the ovary during ovum pick-up, e.g., endometriomas or teratomas measuring >10 mm
5. Has unilateral or bilateral hydrosalpinx that communicates with the endometrial cavity on screening ultrasound or hysterosalpingography.
6. Has intramural fibroids ≥3 cm or submucosal fibroids of any size
7. Has Asherman's syndrome (untreated) or endometrial polyps that have not been resected
8. Has any congenital uterine abnormality which is associated with a decreased chance of pregnancy
9. Inadequate visualization of 1 or both ovaries
10. One or both ovaries not accessible for oocyte retrieval
11. Has a history of recurrent pregnancy losses (i.e., >3 pregnancy losses)
12. Has a history or current evidence of human immunodeficiency virus (HIV) Note: Results obtained within 1 year prior to signing the informed consent form are considered valid.
13. Has tumors of the ovary, breast, uterus, pituitary, or hypothalamus
14. Has a history of epilepsy, thrombophilia, diabetes, untreated or inadequately treated subclinical hypothyroidism, clinically significant cardiovascular, gastrointestinal, hepatic, renal, pulmonary, or auto-immune disease requiring treatment within the last 3 years
15. Is a current smoker who smokes ≥5 cigarettes per day
16. Is assessed by the Investigator as unlikely or unable to adhere to dose and/or visit schedules

Ages: 37 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Fertilized oocyte percentage | Through study completion, an average of 1 year.
  The primary outcome measure will be percentage of fertilized oocytes reaching the blastocyst stage (day 5 or 6 in culture)

SECONDARY OUTCOMES:
coQ10 level | through study completion, an average of 1 year
  CoQ10 levels in plasma and follicular fluid
Protein structural change | through study completion, an average of 1 year
  Rate of structural changes occurring in proteins of the follicular fluid and granulosa (GC) or cumulus (CC) cells representing oxidative stress
MII oocyte percentage | through study completion, an average of 1 year
  Percentage of MII oocytes per total oocytes retrieved, normal 2PN fertilization rate
Reproductive outcome | through study completion, an average of 1 year
  Number of day 3 embryos and ongoing pregnancy rate

CONTACTS AND LOCATIONS:
Locations (1):
- Trio Fertility, Toronto, Ontario, Canada